CLINICAL TRIAL: NCT06509399
Title: Evaluation of the Effectiveness of a Pressure Ulcers Prevention Care Package in the Intensive Care Unit
Brief Title: Care Package for Preventing Pressure Ulcers in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ganime Esra Soysal, Assistant Professor of Surgical Nursing, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SBF-HMS-GES-04
Record Dates: First submitted 2024-06-27; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pressure Ulcer; Nursing Caries
Keywords: Pressure ulcer; Care package; Intensive care unit; Evidence-based practice; Nursing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: experimental study randomised controlled
Who Masked: Participant, Care Provider
Masking Description: The part with patients was completed with a total of 72 patients, 36 in the control group and 36 in the application group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRESSURE ULCERS PREVENTION CARE PACKAGE IN INTENSİVE CARE UNIT (Experimental): This experimental study was carried out in the anesthesia and reanimation intensive care unit of Düzce Atatürk State Hospital. The part with patients was completed with a total of 72 patients, 36 in the control group and 36 in the application group. The occurrence rate of PI was compared between the control group and the application group.
  Interventions: Other: care package
- NURSES' LEVEL OF KNOWLEDGE ABOUT THE CARE PACKAGE (No Intervention): In the section about nurses, no sample was selected and all 50 nurses working in intensive care were included in the study. Nurses' knowledge and attitudes about PI before and after the training were compared.

INTERVENTIONS:
Other: care package — Before the patients in the application group started to be observed, the nurses working in the clinic were trained about the risk assessment, skin assessment, incontinence management, nutrition assessment, positioning, support surfaces and injuries caused by the devices in the BP content to be used in the prevention of IU. After the trainings given to the nurses were completed, care was given to the patients in the practice group in accordance with BP. In addition, patient information was collected from patient information files, nurse observation forms and hospital automation system. In the evaluation step, full compliance with the 7 compliance steps specified in the BP was sought. If any one of these parameters was incomplete, the others were considered as incomplete.
  The patients in the control group were followed up for 30 days until the determined number of patients was reached and their data were collected.
  Arms: PRESSURE ULCERS PREVENTION CARE PACKAGE IN INTENSİVE CARE UNIT

SUMMARY:
The aim of this study is to evaluate the effectiveness of the care package (CP) developed to prevent pressure injury (PI) in patients in intensive care and to evaluate the effect of the training given to nurses on their knowledge levels and attitudes.

DETAILED DESCRIPTION:
This experimental study was carried out in the anesthesia and reanimation intensive care unit of Düzce Atatürk State Hospital. The part with patients was completed with a total of 72 patients, 36 in the control group and 36 in the application group. The occurrence rate of PI was compared between the control group and the application group. In the section about nurses, no sample was selected and all 50 nurses working in intensive care were included in the study. Nurses' knowledge and attitudes about PI before and after the training were compared. Data were analyzed using a statistical program.

ELIGIBILITY:
Inclusion Criteria:

* - 18 years of age or older,
* No development of pressure ulcers in any part of the body,
* Patients expected to stay in the clinic for at least 72 hours or more
* patients with a braden score below 15 points
* Obtaining written consent from the first-degree relatives of patients whose written consent is obtained, patients who are unconscious and unable to give consent

Exclusion Criteria:

* - 18 years of age or younger,
* BY in any part of the body,
* BBYRDS score more than 15
* Failure to give written consent by himself/herself or his/her 1st degree relative
* Exitus, discharge, change of department and the patient's wish to leave the study before completing the number of days determined during the data collection phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Pressure Ulcer Formation | through study completion, an average of 1 year
  Ulcer formation was monitored. Patients were followed up for at least 10 days in this respect.

SECONDARY OUTCOMES:
Knowledge levels of nurses | through study completion, an average of 1 year
  Knowledge levels of nurses were tested before and after the training with the pressure sore assessment form prepared by the researchers.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Abant Izzet Baysal University Faculty of Health Science, Bolu, Merkez
  - Bolu Abant İzzet Baysal Üniversitesi/Sağlık Bilimleri Fakültesi, Bolu

IPD SHARING:
Plan to Share IPD: No